CLINICAL TRIAL: NCT06524466
Title: Neoadjuvant Stereotactic Body Radiotherapy (SBRT) Combined With Lenvatinib and Pucotenlimab for Resectable Hepatocellular Carcinoma With Macrovascular Invasion: A Single-arm, Phase II Study
Brief Title: Neoadjuvant SBRT Combined With Lenvatinib and Pucotenlimab for Resectable Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-694-01
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Resectable Hepatocellular Carcinoma; Macrovascular Invasion; CNLC IIIA Stage
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): After enrollment, patients will immediately begin treatment with Lenvatinib (Len) and Pucotenlimab (Puco). SBRT will be performed within 2-4 weeks after enrollment (with continued Len plus Puco during this period). Six to ten weeks after the completion of SBRT, imaging assessments will be conducted. If there is no sign of tumor progression (PD), surgical resection will be performed within 10-16 weeks after the completion of SBRT. A total of four cycles of Puco treatment must be completed before surgery. The surgical resection should conducted within two weeks after completing the fourth cycle of Puco. Len should be discontinued one week before surgery.
  Interventions: Drug: Neoadjuvant SBRT combined with Lenvatinib and Pucotenlimab

INTERVENTIONS:
Drug: Neoadjuvant SBRT combined with Lenvatinib and Pucotenlimab — SBRT: SBRT will be performed within 2-4 weeks after enrollment. The total radiation dose will be 24 Gy, delivered in 3 fractions on alternate days, to be completed within one week.
  Lenvatinib: 8mg/day, begin immediately after enrollment. Lenvatinib should be discontinued one week before surgery.
  Pucotenlimab: 200mg，3-week interval between cycles, begin immediately after enrollment, a total of four cycles of Puco treatment must be completed before surgery.
  Surgical resection will be performed within 10-16 weeks after the completion of SBRT.

SUMMARY:
At the time of diagnosis, the majority of hepatocellular carcinoma (HCC) patients are at the intermediate to advanced stages, with a 50-70% incidence of macrovascular invasion (including portal vein, hepatic vein, inferior vena cava, or bile duct invasion). Tyrosine kinase inhibitors (TKI, including lenvatinib and sorafenib) or a combination of TKIs and immune therapy is one of the standard treatment options recommended by HCC guidelines. However, numerous retrospective studies have reported that for surgically resectable HCC with macrovascular invasion, surgical resection yields better efficacy than non-surgical treatments (including transarterial interventional therapies and/or systemic therapies). Nevertheless, the postoperative recurrence rate remains exceedingly high, exceeding 80%. Therefore, determining comprehensive approaches to enhance surgical radicality and reduce postoperative recurrence rates is a current research hotspot.

Recent studies have found that neoadjuvant therapy (including immunotherapy alone or in combination with TKI) before surgery can reduce postoperative recurrence rates and extend survival rates. Moreover, SBRT combined with TKI and immunotherapy has a sensitizing effect, particularly showing good sensitivity and control rates for vascular invasion.

Thus, this study aims to conduct a prospective, single-arm phase II clinical trial targeting patients with surgically resectable HCC with macrovascular invasion. The primary endpoints are objective response rate (ORR) and treatment completion rate, to evaluate the efficacy and safety of the preoperative neoadjuvant therapy with the combination of SBRT, lenvatinib, and pucotenlimab (an anti PD-1 drug). The secondary endpoints include progression-free survival (PFS), overall survival (OS), incidence of adverse events, pathological response rate, and incidence of surgical complications, to preliminarily evaluate the efficacy of the neoadjuvant therapy with this triple regimen.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be pathologically confirmed to have hepatocellular carcinoma by biopsy；
2. No previous antitumor treatment;
3. Tumor number ≤ 3, diameter ≤ 10 cm, confined to one lobe of the liver or the middle lobe, evaluated by a surgeon as resectable;
4. Combined with vascular invasion, with the following extents: unilateral portal vein invasion without extending beyond the main portal vein; hepatic vein invasion not reaching the inferior vena cava; unilateral bile duct invasion not reaching the common hepatic duct;
5. No extra-hepatic metastasis or lymph node metastasis.
6. Normal liver volume ≥ 700 cc;
7. Patient KPS ≥ 90;
8. Liver function Child-Pugh class A;
9. Estimated survival of more than 6 months;
10. Function of important organs meets the following requirements: white blood cells ≥ 4.0×10^9/l, neutrophils ≥ 1.5×10^9/l, platelets ≥ 80.0×10^9/l, hemoglobin ≥ 90 g/l; serum albumin ≥ 2.8 g/dl; total bilirubin ≤ 1.5× ULN, ALT/AST/ALP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN or creatinine clearance rate > 60 mL/min; no severe organic diseases;
11. The subject must be able to understand and voluntarily sign a written informed consent form, and must sign the informed consent form prior to any specific procedure of the study, agreeing to comply with the medication and postoperative follow-up requirements as designed in this study.

Exclusion Criteria:

1. Combined with severe impairment of functions of other important organs such as heart, lungs, and kidneys; active infections other than viral hepatitis or other serious comorbid conditions, making the patient unable to tolerate treatment;
2. Diffuse type of HCC, or tumor volume exceeding 50% of liver volume;
3. Portal vein invasion extending beyond the main tract of the portal vein, or hepatic vein invasion reaching the inferior vena cava, or bile duct invasion extending beyond the common hepatic duct;
4. Contraindications to surgical resection, SBRT and immunotherapy;
5. History of other malignant tumors;
6. Combined with immunological diseases or other conditions requiring long-term steroid treatment;
7. Known or suspected allergy to the study drug or any drugs administered in connection with this trial;
8. History of organ transplantation;
9. Pregnant or breastfeeding women;
10. Other factors that may affect patient enrollment and assessment outcomes;
11. Refusal to follow-up according to the requirements set by the study protocol, and refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | From date of neoadjuvant treatment beginning until the date of neoadjuvant treatment completion, up to 1 year.
  The ratio of patients achieving the best efficacy of neoadjuvant therapy, including complete response (CR) and partial response (PR), to all patients.
treatment complete rate (TCR) | From date of neoadjuvant treatment beginning until the date of neoadjuvant treatment completion, up to 1 year.
  The ratio of patients completing the neoadjuvant therapy to all patients.

SECONDARY OUTCOMES:
progression-free survival (PFS) | From date of neoadjuvant treatment beginning until the date of follow-up completion, up to 2 year.
  PFS is defined as the time from treatment to the first confirmed disease progression. For patients who undergo surgical resection, disease progression is defined as postoperative recurrence/metastasis. For patients who do not undergo surgical resection, disease progression is confirmed based on imaging assessment according to the mRECIST criteria.
overall survival (OS) | From date of neoadjuvant treatment beginning until the date of death from any cause, assessed up to 2 years.
  OS is defined as the time from randomization to death from any cause
incidence of adverse events (safety ) | From date of neoadjuvant treatment beginning until 3 months after treatment completion, up to 1 year.
  Treatment-related adverse events are evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0).
perioperative complication rate | The period from the start of surgery to the patient's discharge from hospital, up to 1 year.
  Perioperative complication includes intraoperative complications such as bleeding and transfusion, extensive adhesions, diaphragm resection, prolonged surgery time, etc., as well as postoperative complications such as bleeding, infection, bile leakage, liver dysfunction, etc.
pathological complete response (pCR) | From date of neoadjuvant treatment beginning until the date of surgical resection completion, up to 1 year.
  The ratio of patients with no viable tumor cells in the pathology after resection to all patients undergoing surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Yaojun Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China